CLINICAL TRIAL: NCT05278299
Title: Asia Glaucoma Registry
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof Leung Kai Shun, Christopher, Head and Clinical Professor, The University of Hong Kong
Other Study IDs: UW 21-664
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: POAG

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Glaucoma remains a leading cause for irreversible visual impairment and blindness worldwide and it disproportionately affects people residing in Asia, there is a need to ensure optimal management of the disease in patients with glaucoma. The ability to estimate the rates of structural and functional loss in patients with glaucoma will enable clinicians to identify those with rapidly deteriorating conditions or those at-risk, and to therefore provide timely treatment to these patients. Despite this, there are currently several challenges in identifying rapid-progressors in glaucoma, including lack of consensus on the definition of 'rapid' progression and what rates of change of visual field (VF) encompass clinically significant deterioration relevant to the patients. As such, the Asia Glaucoma Registry is intended to collect data to advance the understanding of glaucoma and its progression in Asia and to understand the management patterns of glaucoma in Asia. The Registry will also provide research data for future collaborative scientific research projects.

DETAILED DESCRIPTION:
Glaucoma remains a leading cause for irreversible visual impairment and blindness worldwide and it disproportionately affects people residing in Asia [Tham et al, 2014]. It is well established that the epidemiology and natural history of glaucoma in patients in the Asia region is different from its western counterparts. Compared with the other parts of the world, the prevalence of primary angle closure glaucoma (PACG) was highest in Asia [Tham et al, 2014]. The prevalence of PACG was higher in East Asia than South East Asia, while the burden of primary open angle glaucoma (POAG) was projected to be the highest in South-Central Asia by 2040 [Chan et al, 2016]; this suggests that ethnic differences within Asia may be a contributing factor to the differences in the prevalence of different types of glaucoma. Furthermore, studies have suggested the prevalence of normal pressure glaucoma is also higher in Asians than Caucasians [ Chen et al , 2020 ] Given the disproportionate burden of glaucoma in Asia, there is a need to ensure optimal management of the disease in patients with glaucoma. The ability to estimate the rates of structural and functional loss in patients with glaucoma will enable clinicians to identify those with rapidly deteriorating conditions or those at-risk, and to therefore provide timely treatment to these patients.

Despite this, there are currently several challenges in identifying rapid-progressors in glaucoma, including lack of consensus on the definition of 'rapid' progression and what rates of change of visual field (VF) encompass clinically significant deterioration relevant to the patients. As such, the Asia Glaucoma Registry is intended to collect data to advance the understanding of glaucoma and its progression in Asia and to understand the management patterns of glaucoma in Asia. The Registry will also provide research data for future collaborative scientific research projects. Glaucoma remains a leading cause for irreversible visual impairment and blindness worldwide and it disproportionately affects people residing in Asia [Tham et al, 2014]. It is well established that the epidemiology and natural history of glaucoma in patients in the Asia region is different from its western counterparts. Compared with the other parts of the world, the prevalence of primary angle closure glaucoma (PACG) was highest in Asia [Tham et al, 2014]. The prevalence of PACG was higher in East Asia than South East Asia, while the burden of primary open angle glaucoma (POAG) was projected to be the highest in South-Central Asia by 2040 [Chan et al, 2016]; this suggests that ethnic differences within Asia may be a contributing factor to the differences in the prevalence of different types of glaucoma. Furthermore, studies have suggested the prevalence of normal pressure glaucoma is also higher in Asians than Caucasians [ Chen et al , 2020 ] Given the disproportionate burden of glaucoma in Asia, there is a need to ensure optimal management of the disease in patients with glaucoma. The ability to estimate the rates of structural and functional loss in patients with glaucoma will enable clinicians to identify those with rapidly deteriorating conditions or those at-risk, and to therefore provide timely treatment to these patients.

Despite this, there are currently several challenges in identifying rapid-progressors in glaucoma, including lack of consensus on the definition of 'rapid' progression and what rates of change of visual field (VF) encompass clinically significant deterioration relevant to the patients. As such, the Asia Glaucoma Registry is intended to collect data to advance the understanding of glaucoma and its progression in Asia and to understand the management patterns of glaucoma in Asia. The Registry will also provide research data for future collaborative scientific research projects.

References:

Chan EW, et al. Glaucoma in Asia: regional prevalence variations and future projections. Br J Opthalmol 2016;100(1):78-85.

Chen MJ. Normal tension glaucoma in Asia : Epidemiology, pathogenesis, diagnosis, and management. Taiwan J Ophthalmo ;10 250-4. He M, et al. Angle-closure glaucoma in East Asian and European people. Different diseases? Eye (Lond) 2006;20(1):3-12.

Tham Y, et al. Global prevalence of glaucoma and projections of glaucoma burden through 2040: a systematic review and metaanalysis. Ophthalmology 2014;121(11):2081-90.

Yip JLY, Foster PJ. Ethnic differences in primary angle-closure glaucoma. Curr Opin Ophthalmol 2006;17(2):175-80.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of POAG or PACG
2. Age ≥18 years at diagnosis.
3. Have reliable VF tests obtained from Humphrey Field Analyzer (HFA) using the same testing strategy on average once a year over 6-7 years backward in at least one eye (the included eye must have evidence of glaucoma as defined above). A reliable VF test has fixation losses ≤20% and false positive errors ≤15%. All criteria mentioned above must be met for inclusion into the study. Both eyes will be included if both eyes meet the inclusion criteria.

Exclusion Criteria:

1. Secondary causes of glaucoma (e.g. uveitic glaucoma, neovascular glaucoma, traumatic glaucoma, exfoliative glaucoma, pigmentary glaucoma, phacomorphic glaucoma, malignant glaucoma)
2. Any neurological disease that may result in VF loss (e.g. stroke)
3. History of optic neuropathy other than glaucoma (including those related to thyroid eye disease);
4. Prior retinal surgery.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A sample size calculation will be conducted to determine the minimum number of subjects to be included in the full-scaled study. Both eyes of patients will be included if both eyes are eligible for inclusion.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of fast progressors among patients with POAG or PACG and the risk factors for fast progression | 1 year

SECONDARY OUTCOMES:
The severity and spectrum of glaucoma in different ethnic groups in Asia and the practice patterns of glaucoma management in Asia | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kai Shun, Christopher Leung, Principal Investigator — The University of Hong Kong
Locations (1):
- Leung Kai Shun, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No